CLINICAL TRIAL: NCT04230291
Title: Evaluating the Effect of a Written Action Plan on Comfort and Understanding of Hidradenitis Suppurativa
Brief Title: Hidradenitis Suppurativa Written Action Plan
Acronym: HSWAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator is not longer at this institution
Sponsor: University of Arizona (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Vivian Shi, MD, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1910019510
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Consultation, then Written Action Plan (Other): CONTROL GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation only
  4. Survey B
  5. Verbal consultation AND Written Action Plan
  6. Survey C
  Interventions: Behavioral: Verbal consultation; Behavioral: Written Action Plan
- Written Action Plan (Experimental): INTERVENTION GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation AND Written Action Plan
  4. Survey C
  Interventions: Behavioral: Written Action Plan

INTERVENTIONS:
Behavioral: Verbal consultation — Verbal consultation only without written information before receiving written action plan
  Arms: Verbal Consultation, then Written Action Plan
Behavioral: Written Action Plan — Written handout of treatment plan and disease management strategies

SUMMARY:
This study is being conducted to evaluate if a written action plan for hidradenitis suppurativa (HS) will help patients with hidradenitis suppurativa gain a better understanding of the condition and how to manage the condition on a daily basis compared to a routine verbal consultation.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of HS

Exclusion Criteria:

* Has been exposed to a written action plan for HS before

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Visits to high-cost care settings | 12 months
  Number of visits to ER, urgent care, or hospitalizations because of HS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No